CLINICAL TRIAL: NCT01453972
Title: Effects of Exercise-intensity on Physiological Adaptations in Overweight and Obese
Acronym: TRENO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRENO
Record Dates: First submitted 2011-10-10; First posted 2011-10-18 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Overweight; Obesity
Keywords: Exercise; High-intensity; Interval training
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Long distanse moderate training (Experimental): 40 minutes moderate treadmill running
  Interventions: Behavioral: Long distanse moderate training
- Long interval training (Experimental): 4x4min interval treadmill running
  Interventions: Behavioral: Long interval training
- Short interval training (Experimental): 10x1min interval treadmill running
  Interventions: Behavioral: Short interval training

INTERVENTIONS:
Behavioral: Long distanse moderate training — Moderate exercise
  Arms: Long distanse moderate training
Behavioral: Long interval training — High-intensity exercise, long duration
  Arms: Long interval training
Behavioral: Short interval training — High intensity exercise, short duration
  Arms: Short interval training

SUMMARY:
The main purpose of our study is to examine the physiological adaptations in oxygen transport chain for high-intensity exercise and moderate exercise in overweight and obese humans. The main goals are:

1. To investigate the most effective short-and long-interval training in terms of VO2max, pulmonary diffusion, cardiac output, endothelial function and mitochondrial function.
2. How these physiological adaptations affect the aerobic endurance and performance, and how this training can reduce the risk of cardiovascular diseases related to overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25

Exclusion Criteria:

* Exclusion criteria will be cardiovascular disease or another disease that is not consistent with high physical activity. Subjects should not have exercised regularly before the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | 6 weeks
  Change in maximal oxygen uptake will be measured after six weeks of various exercise training and related to changes in blood volume, cardiac function, endothelial function and mitochondrial function.

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Medical Faculty, Norwegian University of Science and Technology, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Baekkerud FH, Solberg F, Leinan IM, Wisloff U, Karlsen T, Rognmo O. Comparison of Three Popular Exercise Modalities on V O2max in Overweight and Obese. Med Sci Sports Exerc. 2016 Mar;48(3):491-8. doi: 10.1249/MSS.0000000000000777. PMID 26440134